CLINICAL TRIAL: NCT00426478
Title: The Comparison of the Antihypertensive Efficacy and Tolerability Between Valsartan Plus Hydrochlorothiazide 80mg/12.5mg and Amlodipine 5mg in the Essential Hypertensive Patients
Brief Title: Safety and Efficacy of Valsartan Plus Hydrochlorothiazide and Amlodipine in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631BTW02
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Hypertension
Keywords: AMPM, SBP, DBP, Valsartan plus Hydrochlorothiazide, Amlodipine, high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide; Amlodipine

INTERVENTIONS:
Drug: Valsartan plus Hydrochlorothiazide (80mg/12.5mg)
Drug: Amlodipine (5mg)

SUMMARY:
A double-blind, active-controlled, randomized trial to compare Valsartan plus Hydrochlorothiazide 80mg/12.5mg and Amlodipine 5 mg.

Study design: 2 weeks washout, 8 weeks treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient with age ≧ 18 years old.
* Patient with mild to moderate uncomplicated essential hypertension, and the blood pressure not adequately controlled on existing antihypertensive treatment.
* Patient with sitting systolic blood pressure (sSBP)/ sitting diastolic blood pressure (sDBP) ≦ 180/110 mmHg at screening visit.
* For non-diabetic patient, sitting systolic blood pressure (sSBP) ≧ 140 mmHg or sitting diastolic blood pressure (sDBP) ≧ 90 mmHg at baseline visit; for diabetic patient, sitting systolic blood pressure (sSBP) ≧ 130 mmHg or sitting diastolic blood pressure (sDBP) ≧ 80 mmHg at baseline visit.
* Patient or his/her legally acceptable representative has signed and dated the informed consent form.

Exclusion Criteria:

* Known or suspected secondary hypertension.
* sSBP > 180 mmHg or sDBP > 110 mmHg at baseline visit.
* Patients taking more than two anti-hypertensive medications at the screening visit. (Fixed-dose combinations of two or more antihypertensive therapies will be counted as two or more antihypertensive medications.)
* Known NYHA functional class Chronic Heart Failure (CHF) III and IV.
* With a history of myocardial infarction, transient ischemic attack or cerebrovascular accident within the preceding 6 months, clinically significant valvular heart disease, or hepatic and/or renal dysfunction as defined by the following laboratory parameters
* SGPT (ALT) or SGOT (AST) > two times upper the limit of normal range
* Serum creatinine > 2.3 mg/dl or creatinine clearance < 30 ml/min

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure (msSBP) after 8 weeks treatment

SECONDARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure (msDBP) after 8 weeks treatment
Change from baseline in Ambulatory Blood Pressure Measurement (ABPM) parameters after 8 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah CHAO, MD, Principal Investigator — National Taiwan Univ
Locations (1):
- National Taiwan University, Taipei, R.o.c, Taiwan